CLINICAL TRIAL: NCT01917149
Title: Efficacy and Safety Study of Supramaximal Titrated Inhibition of RAAS in Idiopathic Dilated Cardiomyopathy
Brief Title: Supramaximal Titrated Inhibition of RAAS in Dilated Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Hezheng, Professor, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIRAAS-DC
Record Dates: First submitted 2013-07-30; First posted 2013-08-06 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Dilated Cardiomyopathy
Keywords: Dilated cardiomyopathy; High dose ACEI/ARB
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — benazepril; Valsartan; Metoprolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Metoprolol (Experimental): Patients in the metoprolol group were started on 11.875-23.75mg of metoprolol succinct extended-release tablet once daily (11.875mg was recommended for patients with NYHA functional classes III-IV), and then doses were doubled every 2 weeks to achieve asymptomatic bradycardia (50-60 bpm of heart rate) over 4-6 weeks. Investigators were encouraged to up-titrate metoprolol to a maximum dose of 190mg whenever possible.
  Interventions: Drug: Metoprolol
- Low-dose valsartan (Experimental): Patients randomized to low dose valsartan receive valsartan 80 mg until study completion.
  Interventions: Drug: Valsartan
- Low dose Benazepril (Experimental): Patients randomized to low dose Benazepril receive Benazepril 10 mg until study completion.
  Interventions: Drug: Benazepril
- High dose valsartan (Experimental): Patients randomized to high-dose valsartan were started on valsartan 80mg twice daily, and uptitrated to target doses within 7 days under in-hospital observation. The target high doses of valsartan is determined by left-ventricular end-diastolic diameter (LVEDD) (the maximal value of anteroposterior and lateral diameters) obtained by ECG at the randomization visit. A target dose of valsartan 320mg, 480mg, 640mg daily were assigned to patients with LVEDD of 50-59, 60-69, ≥70 mm respectively.
  Interventions: Drug: Valsartan
- High dose Benazepril (Experimental): Patients randomized to high-dose benazepril were started on benazepril 10mg twice daily, and uptitrated to target doses within 7 days under in-hospital observation. The target high doses of benazepril is determined by left-ventricular end-diastolic diameter (LVEDD) (the maximal value of anteroposterior and lateral diameters) obtained by ECG at the randomization visit. A target dose of benazepril 40mg, 60mg, 80mg daily were assigned to patients with LVEDD of 50-59, 60-69, ≥70 mm respectively.
  Interventions: Drug: Benazepril

INTERVENTIONS:
Drug: Benazepril
  Arms: High dose Benazepril; Low dose Benazepril
Drug: Valsartan
  Arms: High dose valsartan; Low-dose valsartan
Drug: Metoprolol
  Arms: Metoprolol

SUMMARY:
Dilated cardiomyopathy (DCM) is a poorly understood cause of systolic heart failure and is the most common indication for heart transplantation worldwide. Despite advances in medical and device therapy, the 5-year mortality of patients with DCM remains high.

Patients diagnosed of dilated cardiomyopathy with a NYHA functional class of II to IV and left ventricular ejection fraction(LVEF) <35% were selected for randomized controlled study of the efficacy and safety of high dose Renin-angiotensin system (RAS) inhibitor (benazepril or valsartan), in comparison with low dose RAS inhibitor(benazepril or valsartan) and standard beta-adrenergic blocker therapy (metoprolol). The primary endpoint was all cause death or admission for heart failure. Additional prespecified outcomes included all-cause death, cardiovascular death, all-cause admission, heart failure admission. Secondary cardiovascular outcomes included the changes from baseline to the last available observation after treatment in NYHA functional class, quality-of-life scores, LVEF, LVEDD, mitral regurgitation and wall-motion score index assessed by ECG. Adverse events were reported during in-hospital observation and follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dilated cardiomyopathy
* Left ventricular ejection fraction < 35%
* NYHA Functional classes of II-IV
* Symptomatic but not rapidly deteriorating 1 month before enrollment
* Signed informed consent

Exclusion Criteria:

* Contradictions and intolerance of the studied drugs:

  * supine systolic arterial blood pressure < 90 mmHg,
  * renal artery stenosis >50%,
  * pregnancy or lactation,
  * impaired renal function (estimated glomerular filtration rate < 60 ml/min/1.73m2,
  * impaired liver function (total bilirubin >2 times upper limit of normal,
  * serum aspartate AST or alanine ALT >3 times the upper limit of normal),
  * hemoglobin less than 8 mg/dl, hyperkalaemia (serum potassium >5.5mmol/l),
  * obstructive lung disease,
  * advanced atrioventricular block,
  * any co-morbidity with impact on survival, and
  * known intolerance to benazepril, valsartan and metoprolol succinate;
* HF secondary to a known cause:

  * coronary artery disease based on coronary angiography (≥50% stenosis in ≥1 of the major coronary arteries) and/or a history of myocardial infarction or angina pectoris,
  * acute or subacute stage of myocarditis,
  * primary valve disease,
  * diabetes mellitus,
  * excessive use of alcohol or illicit drugs;
* Expected or performed cardiac resynchronization therapy and heart transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2005-03; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
All cause death or admission for heart failure | 48 months after enrollment
  Admission for heart failure was defined as a minimum of 24 h inpatient admission to any health-care facility, with the primary cause being treated for worsening heart failure and during which an additional diuretic drug, intravenous or oral nitrate, or intravenous inotropic agent was given.

SECONDARY OUTCOMES:
Changes in NYHA functional class | 6,12, 24 and 36 months after enrollment
Left-ventricular ejection fraction | 6,12, 24 and 36 months after enrollment
  Left ventricular ejection fraction (LVEF) were calculated from measurements of left ventricular end diastolic and end systolic volumes in apical 4 and 2 chamber views using the modified Simpson's rule according to current guidelines
Left-ventricular end-diastolic diameter | 6, 12 , 24 and 36 months after enrollment

OTHER OUTCOMES:
All-cause mortality | 48 months after enrollment
Cardiovascular death | 48 months after enrollment
All-cause hospital admission | 48 months after enrollment
Heart failure admission | 48 months after enrollment
changes in mitral regurgitation | 12, 24 and 36 months after enrollment
wall-motion score index | 12, 24 and 36 months after enrollment
  Wall motion score index (WMSI) was analyzed using an 11 segments model (3) (basal lateral, middle lateral, basal inferior, middle inferior, basal posterior interventricular septum, middle posterior interventricular septum, basal anterior free wall, middle anterior free wall, basal anterior interventricular septum, middle anterior interventricular septum and apex) with six segments each assigned to anterior and inferior regions, the apex being common. The motion of individual segments was graded as follows: normal 0, hypokinesia 1, akinesia 2, and dyskinesia 3. Global systolic wall motion score was calculated by dividing the total score by the number of segments analyzable. Results were only included when at least four segments from each of the anterior and inferior regions were analyzable. The lowest value of segment motion was chosen from the recorded motion amplitude of all 11 segments
Adverse events | 48 months after enrollment
  Hypotension Hyperkalaemia Renal impairment Liver dysfunction Nonfatal stroke Angioedema

CONTACTS AND LOCATIONS:
Overall Officials: Zheng He, MD, phD, Principal Investigator — Department of Cardiology, Xijing Hospital, Fourth Military Medical University; Qiujun Yu, MD, phD, Principal Investigator — Department of Cardiology, Xijing Hospital, Fourth Military Medical University
Locations (1):
- Xijing Hospital, Department of Cardiology, Xi'an, China

REFERENCES:
- [Derived] He Z, Sun Y, Gao H, Zhang J, Lu Y, Feng J, Su H, Zeng C, Lv A, Cheng K, Li Y, Li H, Luan R, Wang L, Yu Q. Efficacy and safety of supramaximal titrated inhibition of renin-angiotensin-aldosterone system in idiopathic dilated cardiomyopathy. ESC Heart Fail. 2015 Dec;2(4):129-138. doi: 10.1002/ehf2.12042. Epub 2015 Jul 14. PMID 28834619